CLINICAL TRIAL: NCT05800951
Title: Can Escalation Reduce Acute Myocardial Infarction Mortality in Cardiogenic Shock (CERAMICS Study)
Brief Title: Can Escalation Reduce Acute Myocardial Infarction Mortality in Cardiogenic Shock
Acronym: CERAMICS
Status: Enrolling by invitation | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Abiomed Inc. (Industry)
Responsible Party: Principal Investigator, Mir Babar Basir, Director of the Acute Mechanical Circulatory Support Program and STEMI Programs, Henry Ford Health System
Other Study IDs: CERAMICS
Record Dates: First submitted 2022-12-05; First posted 2023-04-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cardiogenic Shock; Acute Myocardial Infarction; STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI; STEMI; NSTEMI; Acute Myocardial Infarction of Right Ventricle (Disorder); Acute Myocardial Infarction of Left Ventricle; Acute Myocardial Infarction With ST Elevation
MeSH Terms: conditions — Shock, Cardiogenic; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CERAMICS study is designed to more clearly delineate the current care of acute myocardial infarction with cardiogenic shock (AMICS) patients who are treated with mechanical circulatory support (MCS) devices in the United States with significant experience in MCS, all of whom have the capability of MCS escalation on-site. Study enrollment is targeted at 120 patients at 20 hospital sites, evaluating clinical outcomes, and focusing on outcomes MCS escalation decision making and ICU level management.

DETAILED DESCRIPTION:
The National Cardiogenic Shock Initiative (NCSI) was an initial step in helping to provide team based protocolized care in AMICS. Over the past 5 years, further evaluation and research has helped identify additional best practices that may contribute to further improving outcomes.

Vasopressors have been identified as being independently associated with worse outcomes and MCS escalation may lead to improvement. While sites participating in the NCSI were early adopters of MCS in AMICS, MCS escalation was open ended and dictated by variable local practice patterns. This contributed to the overall low rate of MCS escalation which occurred in NCSI.

Approximately 30-40% of patients with AMICS have concomitant right ventricular failure (RVF), which is associated with worse morality and may therefore benefit from consideration of early right ventricular mechanical circulatory support (RV-MCS) devices.

A total of 20 total sites will be accepted into the CERAMICS study with the goal of gathering data and outcomes of 120 patients treated at participating centers. The study is expected to collect data for approximately 2 years. Prior to joining the study, each site must have broad adoption of the NCSI treatment algorithm as the standard of care for AMICS among at least 80% of the interventional cardiologists who take STEMI call, as confirmed by the site principal investigator (PI).

It is critically important to track consecutive AMICS patients at each site to assess outcomes by identifying the total sample size treated and to help identify if there were particular biases regarding the use of MCS or escalation of MCS. We will also track survival to hospital discharge of those AMICS patients not treated with MCS via an exclusion form, as well as with patients treated with MCS including when care deviates from the study protocol.

All study data collection is occurring retrospectively at each time-point only using EMR, and there will be no contact between study personnel and patients. Patients will be discharged or deceased at the time of study entry. During participation in the study, study sites will regularly screen all acute MI patient records (STEMI and NSTEMI) for patients who presented with cardiogenic shock (AMICS) via a screening form.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute AMI confirmed by a medical professional, with changes in serum biomarkers or evidence of ischemic EKG changes (STEMI or NSTEMI).
2. Cardiogenic Shock present as defined by the presence of 2 OR MORE of the following criteria prior to PCI:

   * Hypotension: systolic blood pressure ≤ 90mmHg at baseline (prior to PCI) or the use of inotropes or vasopressors to maintain SBP ≥ 90mmHg
   * Evidence of end organ hypoperfusion: elevated serum lactate levels (venous or arterial), cool extremities, oliguria/anuria
   * Hemodynamic criteria: Cardiac Index of < 2.2 L/min/m2 or a cardiac power output (CPO) of ≤ 0.6 watts
3. Patient underwent PCI within 12 hours of hospital presentation.

Exclusion Registry Exclusion Criteria:

AMICS patients who meet any of the following study exclusion criteria will have a limited set of data collected via a single-page Patient Exclusion Form completed and submitted within 45 days of hospital discharge, which includes the reason for exclusion, date of index PCI, and assessment of patient survival to hospital discharge:

1. Evidence of Anoxic Brain Injury
2. Unwitnessed out of hospital cardiac arrest or any cardiac arrest in which return of spontaneous circulation (ROSC) is not achieved within 30 minutes
3. IABP placed prior to MCS
4. Septic, anaphylactic, hemorrhagic, and neurologic causes of shock
5. Non-ischemic causes of shock/hypotension (pulmonary embolism, pneumothorax, myocarditis, tamponade, etc.)
6. Active bleeding for which MCS is contraindicated
7. Recent major surgery for which MCS is contraindicated
8. Mechanical complications of AMI (acute ventricular septal defect (VSD) or acute papillary muscle rupture)
9. Known left ventricular thrombus for which MCS is contraindicated
10. Mechanical aortic prosthetic valve
11. Contraindication to intravenous systemic anticoagulation which precludes placement of MCS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present with an acute myocardial infarction (AMI) with cardiogenic shock (AMICS) prior to PCI.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital discharge survival/survival at 30 days | Hospital discharge survival/survival at 30 days
  Hospital discharge survival/survival at 30 days

SECONDARY OUTCOMES:
All-cause mortality at 1 year | All-cause mortality at 1 year
  All-cause mortality at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mir B Basir, DO, Principal Investigator — Henry Ford Health; William W O'Neill, MD, Principal Investigator — Henry Ford Health
Locations (17):
- United States (17):
  - Loma Linda University Medical Center, Loma Linda, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Providence St. Joseph Hospital Orange, Orange, California
  - St. Anthony Hospital, Lakewood, Colorado
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Northside Hospital Atlanta, Atlanta, Georgia
  - St. Elizabeth Edgewood Hospital, Edgewood, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Ascenion St. John Hospital, Detroit, Michigan
  - Spectrum Health Hospitals Fred and Lena Meijer Heart Center, Grand Rapids, Michigan
  - Hackensack Meridian Jersey Shore University Medical Center, Neptune City, New Jersey
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Parkwest Medical Center, Nashville, Tennessee
  - Methodist Hospital, San Antonio, Texas
  - UVA University Hospital, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basir MB, Schreiber T, Dixon S, Alaswad K, Patel K, Almany S, Khandelwal A, Hanson I, George A, Ashbrook M, Blank N, Abdelsalam M, Sareen N, Timmis SBH, O'Neill Md WW. Feasibility of early mechanical circulatory support in acute myocardial infarction complicated by cardiogenic shock: The Detroit cardiogenic shock initiative. Catheter Cardiovasc Interv. 2018 Feb 15;91(3):454-461. doi: 10.1002/ccd.27427. Epub 2017 Dec 20. PMID 29266676
- [Background] Hanson ID, Tagami T, Mando R, Kara Balla A, Dixon SR, Timmis S, Almany S, Naidu SS, Baran D, Lemor A, Gorgis S, O'Neill W, Basir MB; National Cardiogenic Shock Investigators. SCAI shock classification in acute myocardial infarction: Insights from the National Cardiogenic Shock Initiative. Catheter Cardiovasc Interv. 2020 Nov;96(6):1137-1142. doi: 10.1002/ccd.29139. Epub 2020 Jul 16. PMID 32672388
- [Background] Goldsweig AM, Tak HJ, Alraies MC, Park J, Smith C, Baker J, Lin L, Patel N, O'Neill WW, Basir MB; National Cardiogenic Shock Initiative Investigators. Mechanical Circulatory Support Following Out-of-Hospital Cardiac Arrest: Insights From the National Cardiogenic Shock Initiative. Cardiovasc Revasc Med. 2021 Nov;32:58-62. doi: 10.1016/j.carrev.2020.12.021. Epub 2020 Dec 23. PMID 33358390
- [Background] Lemor A, Basir MB, Gorgis S, Todd J, Marso S, Gelormini J, Akhtar Y, Baker J, Chahin J, Abdul-Waheed M, Thukral N, O'Neill W. Impact of Age in Acute Myocardial Infarction Cardiogenic Shock: Insights From the National Cardiogenic Shock Initiative. Crit Pathw Cardiol. 2021 Sep 1;20(3):163-167. doi: 10.1097/HPC.0000000000000255. PMID 33606413
- [Background] Basir MB, Kapur NK, Patel K, Salam MA, Schreiber T, Kaki A, Hanson I, Almany S, Timmis S, Dixon S, Kolski B, Todd J, Senter S, Marso S, Lasorda D, Wilkins C, Lalonde T, Attallah A, Larkin T, Dupont A, Marshall J, Patel N, Overly T, Green M, Tehrani B, Truesdell AG, Sharma R, Akhtar Y, McRae T 3rd, O'Neill B, Finley J, Rahman A, Foster M, Askari R, Goldsweig A, Martin S, Bharadwaj A, Khuddus M, Caputo C, Korpas D, Cawich I, McAllister D, Blank N, Alraies MC, Fisher R, Khandelwal A, Alaswad K, Lemor A, Johnson T, Hacala M, O'Neill WW; National Cardiogenic Shock Initiative Investigators. Improved Outcomes Associated with the use of Shock Protocols: Updates from the National Cardiogenic Shock Initiative. Catheter Cardiovasc Interv. 2019 Jun 1;93(7):1173-1183. doi: 10.1002/ccd.28307. Epub 2019 Apr 25. PMID 31025538
- [Background] Ahlers MJ, Srivastava PK, Basir MB, O'Neill WW, Hacala M, Ammar K, Khalil S, Hollowed J, Nsair A. Characteristics and outcomes of patients presenting with acute myocardial infarction and cardiogenic shock during COVID-19. Catheter Cardiovasc Interv. 2022 Oct;100(4):568-574. doi: 10.1002/ccd.30390. Epub 2022 Sep 7. PMID 36073018
- See also: Henry Ford Hospital web page for NCSI/CERAMICS — https://www.henryford.com/cardiogenicshock

DOCUMENTS (1):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT05800951/Prot_000.pdf